CLINICAL TRIAL: NCT01528449
Title: Blood Donation Screening for Babesia Microti by Real-time Polymerase Chain Reaction (PCR) and by Indirect Flourescent Antibody (IFA) Assays
Brief Title: Babesia Testing in Blood Donors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imugen (Industry)
Collaborators: American National Red Cross (Other); Memorial Blood Centers, Minnesota (Other); Rhode Island Blood Center (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BNATIFA-10; NCT01525030 (obsolete NCT alias)
Record Dates: First submitted 2012-01-31; First posted 2012-02-08 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Transfusion Transmitted Babesiosis
Keywords: babesia; blood donation; transfusion transmitted babesiosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- retrospective (Experimental): archived specimens from blood donors whose units have already been released and transfused into recipients will be tested. Attempts will be made to contact and obtain follow up specimens from both the donor and recipient of units initially testing positive for B.microti. the interventions are investigational diagnostic tests for B.microti (PCR and IFA).
  Interventions: Biological: B.microti diagnostic blood tests
- prospective, real time (Experimental): specimens from current blood donors will be tested and those testing positive for B.microti will not be released and the units will be disgarded, and the donors notified and deferred from future blood donation. the interventions are investigational diagnostic tests for B.microti (PCR and IFA).
  Interventions: Biological: B.microti diagnostic blood tests

INTERVENTIONS:
Biological: B.microti diagnostic blood tests — the interventions/procedures are investigational diagnostic tests for B.microti (PCR and IFA).
  Other Names: proprietary in-house developed PCR and IFA Babesia doagnostic tests
  Arms: retrospective
Biological: B.microti diagnostic blood tests — the interventions/procedures are investigational diagnostic tests for B.microti (PCR and IFA).
  Arms: prospective, real time

SUMMARY:
Both prospective and retrospective (look back) study of blood donors for laboratory evidence of babesia microti infection.

Two laboratory methodologies will be utilized:

1. - PCR, to look for the presence of B.microti in whole blood
2. - IFA, to look for significant titers of B.microti antibody

DETAILED DESCRIPTION:
Retrospective study will involve archived specimens from blood donors whose units have already been released and transfused into recipients.

Prospective study will be real time and units testing positive by either PCR or IFA will be not released and will be disgarded, and the donors advised and deferred from further blood donation

ELIGIBILITY:
Inclusion Criteria:

* same as for donating blood

Exclusion Criteria:

* donor refusual to sign informed consent for this investigational babesia testing

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90116 (Actual)
Dates: Start 2011-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
number of blood donors testing positive for evidence of Babesia infection | goal is up to one year (all specimens by end 2012)

SECONDARY OUTCOMES:
the number of cases of transfusion transmitted babesia infection identified | goal is up to one year (all specimens by end 2012)

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Molloy, MD, Principal Investigator — Imugen Medical Director
Locations (1):
- Imugen, Norwood, Massachusetts, United States

REFERENCES:
- [Derived] Moritz ED, Winton CS, Tonnetti L, Townsend RL, Berardi VP, Hewins ME, Weeks KE, Dodd RY, Stramer SL. Screening for Babesia microti in the U.S. Blood Supply. N Engl J Med. 2016 Dec 8;375(23):2236-2245. doi: 10.1056/NEJMoa1600897. PMID 27959685